CLINICAL TRIAL: NCT00308282
Title: Phase II Study of Safety and Efficacy of Intravenous LY2127399 in Patients With Rheumatoid Arthritis Treated With Methotrexate
Brief Title: A Multi-Site Study to Evaluate the Safety and Effect of Study Drug on Participants With Rheumatoid Arthritis
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Eli Lilly and Company (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: 11055; H9B-MC-BCDF (Other: Eli Lilly and Company)
Record Dates: First submitted 2006-03-28; First posted 2006-03-29 (Estimated); Results first posted 2019-03-18 (Actual); Last update posted 2019-09-10 (Actual); Status verified 2019-08

CONDITIONS: Arthritis, Rheumatoid
MeSH Terms: conditions — Arthritis, Rheumatoid | interventions — tabalumab

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- A (Experimental)
  Interventions: Drug: LY2127399
- B (Placebo Comparator)
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: LY2127399 — 30 mg, 60 mg or 160 mg, IV (in the vein) in weeks 0, 3 and 6. Treatment duration: 6 weeks.
  Arms: A
Drug: Placebo — IV (in vein) in weeks 0, 3 and 6. Treatment duration: 6 weeks.
  Arms: B

SUMMARY:
This study is a multicenter, double-blind, study to evaluate the safety and effectiveness of treatment with LY2127399 (in addition to the standard of care treatment, methotrexate) for participants with Rheumatoid Arthritis. Participants will receive three intravenous doses of LY2127399 or placebo. Participants will participate in 10 or more visits to the study site, over 6 months. Evaluation of safety and efficacy will be conducted throughout the study.

ELIGIBILITY:
Inclusion Criteria:

* Male or female between the ages of 18 and 75 years
* Have given written informed consent approval
* Women must not be at risk to become pregnant during study participation
* Diagnosis of Rheumatoid Arthritis according to the 1987 revised American Rheumatism Association (ARA) criteria for the classification of RA
* Serum C-reactive protein (CRP) measurement greater than the upper limit of normal (ULN, 0.574 mg/dL), or erythrocyte sedimentation rate (ESR) ≥28 mm/hr
* Current, regular use of Methotrexate, at a stable dose
* Biologic DMARD naïve, and have had an insufficient response (in the opinion of the investigator) to an adequate therapeutic dose of at least 1 oral DMARD

Exclusion Criteria:

* Use of excluded medications (reviewed by study doctor)
* Surgical treatment of a joint with 2 months of study enrollment that is to be assessed in the study
* Are unable to ambulate; that is, confined to bed or wheelchair bound
* Have medical findings which, in the opinion of the study doctor, put participant at an unacceptable risk for participation in the study
* Have had recent or ongoing infection which, in the opinion of the study doctor put participant at an unacceptable risk for participation.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 136 (Actual)
Dates: Start 2006-03-28 (Actual); Primary Completion 2007-06-18 (Actual); Study Completion 2007-10-18 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Call 1-877-CTLILLY (1-877-285-4559) or 1-317-615-4559 Mon - Fri 9 AM - 5 PM Eastern time (UTC/GMT - 5 hours, EST), Study Director — Eli Lilly and Company
Locations (14):
- Romania (14):
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Bacau
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Baia Mare
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Brasov
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Brăila
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Bucharest
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Cluj-Napoca
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Constanța
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Craiova
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Iași
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Sf. Gheorghe
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Sibiu
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Târgovişte
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Târgu Mureş
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Timișoara

IPD SHARING:
Plan to Share IPD: Yes
Anonymized individual patient level data will be provided in a secure access environment upon approval of a research proposal and a signed data sharing agreement.
Supporting Information: Study Protocol, SAP, CSR
Time Frame: Data are available 6 months after the primary publication and approval of the indication studied in the US and EU, whichever is later. Data will be indefinitely available for requesting.
Access Criteria: A research proposal must be approved by an independent review panel and researchers must sign a data sharing agreement.
URL: https://vivli.org/

REFERENCES:
- [Derived] Genovese MC, Bojin S, Biagini IM, Mociran E, Cristei D, Mirea G, Georgescu L, Sloan-Lancaster J. Tabalumab in rheumatoid arthritis patients with an inadequate response to methotrexate and naive to biologic therapy: a phase II, randomized, placebo-controlled trial. Arthritis Rheum. 2013 Apr;65(4):880-9. doi: 10.1002/art.37820. PMID 23359344
- See also: Lilly Clinical Trial Registry — http://www.lillytrials.com

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Study populations are based on randomized treatment groups. Safety and Pharmacokinetic (PK) populations were adjusted due to dosing errors and account for actual treatment received.
Pre-assignment Details: Completers were defined as having completed 3 infusions and required follow-up visits.
Groups:
- Placebo: Placebo administered IV in weeks 0, 3 and 6. Treatment duration: 6 weeks.
- 30 mg LY2127399: 30 milligram (mg) LY2127399 administered Intravenously (IV) in weeks 0, 3 and 6. Treatment duration: 6 weeks.
- 60 mg LY2127399: 60 mg LY2127399 administered Intravenously (IV) in weeks 0, 3 and 6. Treatment duration: 6 weeks.
- 160 mg LY2127399: 160 mg LY2127399 administered Intravenously (IV) in weeks 0, 3 and 6. Treatment duration: 6 weeks.
Period: Overall Study
Arm/Group | Placebo | 30 mg LY2127399 | 60 mg LY2127399 | 160 mg LY2127399
Started | 34 | 34 | 34 | 34
Received at Least One Dose of Study Drug | 34 | 34 | 34 | 34
Completed | 31 | 30 | 33 | 32
Not Completed | 3 | 4 | 1 | 2

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Placebo | 30 mg LY2127399 | 60 mg LY2127399 | 160 mg LY2127399 | Total
Number analyzed (Participants) | 34 | 34 | 34 | 34 | 136
Age, Customized [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0 | 0 | 0
  Between 18 and 73 years | 34 | 34 | 34 | 34 | 136
  >=73 years | 0 | 0 | 0 | 0 | 0
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 29 | 31 | 26 | 29 | 115
  Male | 5 | 3 | 8 | 5 | 21
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0 | 0 | 0 | 0 | 0
  Not Hispanic or Latino | 34 | 34 | 34 | 34 | 136
  Unknown or Not Reported | 0 | 0 | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0 | 0 | 0
  Asian | 0 | 0 | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0 | 0 | 0
  Black or African American | 0 | 0 | 0 | 0 | 0
  White | 34 | 34 | 34 | 34 | 136
  More than one race | 0 | 0 | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0 | 0 | 0
ACR functional class [Count of Participants; unit: Participants] — ACR American College of Rheumatology.
  Class I: Completely able to perform usual activities of daily living (self-care, vocational, and avocational).
  Class II: Able to perform usual self-care and vocational activities (work, school, homemaking), but limited in avocational activities (recreation and/or leisure).
  Class III: Able to perform usual self-care activities, but limited in vocational and avocational activities.
  Class IV: Limited in availability to perform usual self-care, vocational, and avocational activities.
  Participants
    Class I | 4 | 4 | 3 | 7 | 18
    Class II | 15 | 19 | 19 | 16 | 69
    Class III | 15 | 11 | 12 | 11 | 49

OUTCOME MEASURES:

1. Primary Outcome: Percentage of Participants Achieving American College of Rheumatology 20% Response (ACR20) (Effectiveness of LY2127399 in Treating Rheumatoid Arthritis Using the ACR20 Scale)
Description: ACR Responder Index is a Composite of clinical, laboratory, and functional measures of rheumatoid arthritis (RA). ACR20 Responders: had ≥20% improvement from baseline in both tender and swollen joint counts and ≥20% improvement in at least 3 of 5 criteria: participant's and physician's global assessment of disease activity, Health Assessment Questionnaire-Disability Index (HAQ-DI) (which measured participants' perceived degree of difficulty performing daily activities), visual analog pain scale, and erythrocyte sedimentation rate (ESR) or C-reactive protein (CRP).
Time Frame: Week 16
Population: All participants who received at least 1 dose of study drug who had a baseline and at least 1 post-baseline ACR value.
Measure: Number; unit: percentage of participants
Arm/Group | Placebo | 30 mg LY2127399 | 60 mg LY2127399 | 160 mg LY2127399
Number analyzed (Participants) | 34 | 33 | 34 | 33
percentage of participants | 29.4 | 57.6 | 67.6 | 51.5

2. Secondary Outcome: Number of Participants With Treatment Emergent Adverse Events (TEAE) (Safety of Repeat Doses (3) of LY2127399 Through Evaluation of Laboratory Tests, Vital Signs and Electrocardiograms)
Description: Treatment-emergent adverse events (TEAEs) were defined as those AEs with start date and time equal to or after the start of study medication infusion. In the case of a missing onset time for an AE, an AE with a start date equal to or greater than the dosing date was considered treatment-emergent. A summary of other nonserious AEs, and all SAE's, regardless of causality, is located in the Reported Adverse Events section.
  All participants who received at least one dose of study drug. Due to dosing errors (a participant received 60 mg LY2127399 in the placebo group), the safety population was adjusted to account for actual treatment received.
Time Frame: Baseline through Study Completion (Up to 19 Months)
Population: All participants who received at least one dose of study drug. Due to dosing errors (a participant received 60 mg LY2127399 in the placebo group), the safety population was adjusted to account for actual treatment received.
Measure: Count of Participants; unit: Participants
Arm/Group | Placebo | 30 mg LY2127399 | 60 mg LY2127399 | 160 mg LY2127399
Number analyzed (Participants) | 33 | 34 | 35 | 34
Participants | 15 | 14 | 15 | 15

3. Secondary Outcome: Evaluation of the Pharmacokinetics of LY2127399: Clearance
Description: Population estimate of constant clearance as determined by population PK analysis. A 2-compartment model was used in PK modeling. Constant clearance is the PK parameter which describes the linear elimination of LY2127399 from serum.
Time Frame: 2 hours pre-dose, pre-dose, 1 hour and 4 hour(s) post dose
Population: All participants who received at least one dose of LY2127399 and had evaluable PK data.
Measure: Mean (Standard Deviation); unit: Liters per Hour (L/Hr)
Arm/Group | 30 mg LY2127399 | 60 mg LY2127399 | 160 mg LY2127399
Number analyzed (Participants) | 32 | 31 | 34
Liters per Hour (L/Hr) | 0.0079 (0.0031) | 0.0062 (0.0023) | 0.0054 (0.0021)

4. Secondary Outcome: Percentage of Participants Achieving ACR 50 and ACR70
Description: ACR Responder Index: composite of clinical, laboratory, and functional measures of Rheumatoid Arthritis (RA). ACR50 and ACR70 Responder: had either a ≥50% or ≥70% improvement from baseline in both tender and swollen joint counts and either a ≥50% or ≥70% improvement in at least 3 of 5 criteria: participant's (Pt's) and physician's global assessment of disease activity, HAQ-DI (measured Pts' perceived degree of difficulty performing daily activities), joint pain, and CRP (respectively).
Time Frame: Baseline through Week 24
Population: All participants who received at least 1 dose of study drug who had a baseline and at least 1 post-baseline ACR value.
Measure: Number; unit: percentage of participants
Arm/Group | Placebo | 30 mg LY2127399 | 60 mg LY2127399 | 160 mg LY2127399
Number analyzed (Participants) | 34 | 33 | 34 | 33
percentage of participants
  ACR50 | 20.6 | 57.6 | 55.9 | 42.4
  ACR70 | 2.9 | 24.2 | 17.6 | 9.1

5. Secondary Outcome: Change From Baseline in the Disease Activity Score 28 Joint Count (DAS28-CRP)
Description: Disease Activity Score (DAS) modified to include 28 joint count (DAS28) consisted of composite score of following variables: tender joint count (TJC28), swollen joint count (SJC28), CRP [milligrams per liter (mg/L)], and participant's global assessment of disease activity using visual analog scale (VAS) (participant global VAS). DAS28-CRP=0.56*square root (sqrt)(TJC28)+0.28*sqrt(SJC28)+0.36*natural log(CRP+1)+0.014*participant global VAS+0.96. Scores ranged from 1.0-9.4, where lower scores indicated less disease activity and remission is DAS28-CRP <2.6. A negative change indicated an improvement.
Time Frame: Baseline, Week 24
Population: All participants who received at least 1 dose of study drug who had a baseline and at least 1 post-baseline ACR value.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Placebo | 30 mg LY2127399 | 60 mg LY2127399 | 160 mg LY2127399
Number analyzed (Participants) | 34 | 33 | 34 | 33
units on a scale | -0.78 (0.835) | -1.68 (0.862) | -1.62 (1.007) | -1.46 (0.899)

6. Secondary Outcome: European League Against Rheumatism (EULAR28) Response: Percentage of Participants With Combined Good and Moderate Responses
Description: EULAR Responder index based on 28 joint counts categorizes clinical response based on improvement since baseline in DAS28-CRP. DAS28-CRP scores range from 1.0-9.4, where lower scores indicated less disease activity. High disease activity: DAS28-CRP >5.1, low disease activity: DAS28-CRP <3.2, and remission: DAS28-CRP <2.6. Participants are categorized as EULAR responders or non-responders (NR) based on improvement of DAS28-CRP scores from baseline. EULAR DAS28-CRP responder index defines a good (absolute: <3.2 or >1.2 improvement from baseline), moderate (absolute: 3.2-5.1 or 0.6-1.2 improvement from baseline), or no response (absolute: >5.1 or <0.6 improvement from baseline). Percentage of participants with DAS28-CRP based EULAR response =(number of participants with specific response) / (number of participants analyzed in the group) * 100.
Time Frame: Baseline, Week 24
Population: All participants who received at least 1 dose of study drug who had a baseline and at least 1 post-baseline ACR value.
Measure: Number; unit: percentage of participants
Arm/Group | Placebo | 30 mg LY2127399 | 60 mg LY2127399 | 160 mg LY2127399
Number analyzed (Participants) | 34 | 33 | 34 | 33
percentage of participants | 52.9 | 90.9 | 88.2 | 81.8

7. Secondary Outcome: Change From Baseline (CFB) in Serum Immunoglobulins IgG, IgA and IgM
Description: Immunoglobulins (Ig), or antibodies, are large proteins used by the immune system to identify and neutralize foreign particles such as bacteria and viruses. Their normal blood levels indicate proper immune status. A negative change indicates a decrease in Ig levels.
Time Frame: Baseline, Week 24
Population: All participants who received one dose of study drug and had post baseline serum immunoglobulin data.
Measure: Mean (Standard Deviation); unit: milligrams per deciliter (mg/dL)
Arm/Group | Placebo | 30 mg LY2127399 | 60 mg LY2127399 | 160 mg LY2127399
Number analyzed (Participants) | 32 | 31 | 31 | 33
milligrams per deciliter (mg/dL)
  IgG | 6.2 (141.29) | -26.7 (185.55) | -97.2 (313.71) | -72.0 (163.20)
  IgA | -18.9 (44.00) | -11.1 (42.28) | -27.5 (58.00) | -32.6 (39.71)
  IgM | 1.6 (15.99) | -7.1 (41.76) | -18.6 (55.50) | -29.0 (33.72)

8. Secondary Outcome: Change From Baseline in CD20+ B Cell Number Count
Description: CD20+ B-cells are a disease-related peripheral blood biomarker used to assess disease progression of Rheumatoid Arthritis (RA). A reduction in CD20+ B-cell values may indicate an improvement in RA symptoms.
Time Frame: Baseline, Week 24
Population: All participants who received one dose of study drug and had post baseline CD20+ cell data.
Measure: Mean (Standard Deviation); unit: Cells per microLiter
Arm/Group | Placebo | 30 mg LY2127399 | 60 mg LY2127399 | 160 mg LY2127399
Number analyzed (Participants) | 32 | 31 | 32 | 33
Cells per microLiter | -46.9 (74.51) | -56.3 (84.75) | -135.9 (179.6) | -59.2 (81.31)

ADVERSE EVENTS:
Description: All participants who received at least one dose of study drug. Due to dosing errors (a participant received 60 mg LY2127399 in the placebo group), the safety population was adjusted to account for actual treatment received.
Arm/Group | Placebo | 30 mg LY2127399 | 60 mg LY2127399 | 160 mg LY2127399
Serious Adverse Events (participants affected / at risk) | 3/33 | 2/34 | 0/35 | 3/34
Other Adverse Events (participants affected / at risk) | 15/33 | 14/34 | 15/35 | 15/34
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Placebo (N=33) | 30 mg LY2127399 (N=34) | 60 mg LY2127399 (N=35) | 160 mg LY2127399 (N=34)
Anemia (Blood and lymphatic system disorders) | 1 | 0 | 0 | 0
Gastritis Haemorrhagic (Gastrointestinal disorders) | 1 | 0 | 0 | 0
Bile Duct Stone (Hepatobiliary disorders) | 1 | 0 | 0 | 0
Drug Hypersensitivity (Immune system disorders) | 0 | 1 | 0 | 1
Necrotising Fasciitis (Infections and infestations) | 1 | 0 | 0 | 0
Urinary Tract Infection (Infections and infestations) | 0 | 0 | 0 | 1
Rheumatoid Arthritis (Musculoskeletal and connective tissue disorders) | 0 | 1 | 0 | 0
Endometrial Cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 0 | 1
Hydronephrosis (Renal and urinary disorders) | 0 | 0 | 0 | 1
Pleural Effusion (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 1
OTHER ADVERSE EVENTS (reported when occurring in more than 2% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Placebo (N=33) | 30 mg LY2127399 (N=34) | 60 mg LY2127399 (N=35) | 160 mg LY2127399 (N=34)
Alanine Aminotransferase Increased (Investigations) | 4 | 2 | 3 | 3
Aspartate Aminotransferase Increased (Investigations) | 4 | 2 | 3 | 3
Blood Pressure Increased (Investigations) | 2 | 2 | 1 | 1
Gamma Glutamyl Transferase Increased (Investigations) | 0 | 2 | 1 | 1
Blood Alkaline Phosphatase Increased (Investigations) | 0 | 2 | 1 | 0
Upper respiratory tract infections (Infections and infestations) | 0 | 2 | 0 | 2
Ventricular Extrasystoles (Cardiac disorders) | 0 | 1 | 3 | 2
Myocardial Ischemia (Cardiac disorders) | 0 | 1 | 2 | 0
Abdominal pain upper (Gastrointestinal disorders) | 0 | 3 | 2 | 2
Nausea (Gastrointestinal disorders) | 1 | 2 | 3 | 2
Headache (Nervous system disorders) | 1 | 3 | 2 | 1
Dizziness (Nervous system disorders) | 2 | 1 | 0 | 3
Leukopenia (Blood and lymphatic system disorders) | 2 | 1 | 0 | 2
Back Pain (Musculoskeletal and connective tissue disorders) | 1 | 1 | 1 | 1
Cough (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1 | 0
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1 | 0
Interstitial Lung Disease (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0 | 0
Pharyngolaryngeal Pain (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 1
Pleural Effusion (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0 | 1
Pleurisy (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 1
Rhinorrhoea (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1 | 0
Chills (General disorders) | 0 | 1 | 0 | 0
Injection Site Irritation (General disorders) | 0 | 0 | 0 | 1
Malaise (General disorders) | 1 | 0 | 0 | 0
Pyrexia (General disorders) | 0 | 0 | 0 | 1
Thirst (General disorders) | 0 | 0 | 0 | 1

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of more than 60 days